CLINICAL TRIAL: NCT03151213
Title: Effect of Preoperative Administration of Oral Pregabalin on the Postoperative Analgesia in Patients Scheduled for Radiofrequency Ablationof Focal Lesions in the Liver
Brief Title: Effect of Pregabalin on the Postoperative Analgesia in RFA of Focal Lesions in the Liver
Acronym: pregabalin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, PhDTropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: amr magdy
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double blinded by closed envelops
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin (Active Comparator): Pregabalin 150 mg before intervention
  Interventions: Drug: Pregabalin 150mg
- Placebo (Placebo Comparator): Placebo before intervention
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pregabalin 150mg — Pregabalin 150mg before RFA of liver cancer
  Other Names: pregab
  Arms: Pregabalin
Other: Placebo — Placebo before RFA of liver cancer
  Arms: Placebo

SUMMARY:
The study aimed to investigate the preemptive analgesia efficacy of of preemptive pregabalin for the postoperative pain management after radiofrequency ablation (RFA) of liver cancer.

DETAILED DESCRIPTION:
Our data will investigate if preemptive administration of pregabalin will have a role in reducing postoperative pain after radiofrequency ablation (RFA) of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* HCC patients, Child A, B, scheduled for Radiofrequency ablation of HCC.

Exclusion Criteria:

* Encephalopathy, Renal impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
visual analogue pain scale (VAS Pain) post operatively | 2 weeks
  Amplitude of pain postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Amr Magdy Abdelfattah, consultant, Principal Investigator — Tanta University Faculty of Medicine; Sherief Abd-Elsalam, Consultant, Study Director — Tanta university Faculty of Medicine
Locations (1):
- Tanta university - faculty of medicine, Cairo, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided